CLINICAL TRIAL: NCT02312453
Title: Posterior Parasagittal In-Plane Ultrasound-Guided Infraclavicular Brachial Plexus Block - A Case Series
Brief Title: Posterior Parasagittal In-Plane Ultrasound-Guided Infraclavicular Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Beh Zhi Yuen, Dr, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1038.76
Record Dates: First submitted 2014-11-28; First posted 2014-12-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Brachial Plexus Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Posterior approach (Experimental): All patients were given a single shot ultrasound-guided posterior parasagittal in-plane approach infraclavicular brachial plexus block under aseptic technique. The blocks were performed using a 21G, 100 mm insulated short bevel needle (Stimuplex A, B Braun, Melsungen, Germany) without nerve stimulation. A 25-ml local anaesthetic admixture [Lignocaine 2% (100mg) plus Ropivacaine 0.75% (150mg)] was administered. We used an ultrasound machine (Sonosite M-Turbo; Sonosite®, Bothell, WA, USA) with HFL38x/ 13-6 MHz linear transducer probe.
  Interventions: Procedure: Posterior approach

INTERVENTIONS:
Procedure: Posterior approach — We adopted the technique as described by Hebbard et al.
  Other Names: posterior approach parasagittal in-plane

SUMMARY:
Abstract

Introduction: The brachial plexus at the infraclavicular level runs deeper compared to its course proximally, giving rise to impaired needle visualisation due to the steep angle of needle insertion with the current ultrasound-guided approach. A new posterior parasagittal in-plane ultrasound-guided infraclavicular approach was introduced to improve needle visibility. However no further follow up study was done.

Methods: We performed a case series and a cadaveric dissection to assess its feasibility in a single centre, University of Malaya Medical Centre, Kuala Lumpur, Malaysia from November 2012 to October 2013. After obtaining approval from the Medical Ethics Committee, University Malaya Medical Centre, 18 patients undergoing upper limb surgery were prospectively recruited. A cadaveric dissection was also performed. The endpoints of this study were the success rate, performance time, total anaesthesia related time, quality of anaesthesia and any incidence of complications.

DETAILED DESCRIPTION:
Introduction Our study focus on the ultrasound guided infraclavicular brachial plexus block, which is a cord-level block of the brachial plexus for surgical procedures below mid-humerus. The brachial plexus at this level runs deeper compared to its course proximally, giving rise to impaired needle visualisation due to the steep angle of needle insertion with the current ultrasound-guided approach (lateral para-sagittal in-plane technique).1

A new ultrasound-guided posterior approach parasagittal in-plane infraclavicular block was introduced to improve needle visibility.2 However no further follow up study was done.

Therefore, we performed a case series of 18 patients with a cadaveric dissection, to assess the feasibility of this approach.

Methods After obtaining ethics committee approval from the Medical Ethics Committee, University Malaya Medical Center, Kuala Lumpur, Malaysia (Chairperson Professor Dr. Looi Lai Meng; IRB reference no. 949.14 dated 17 October 2012, amendment no.1038.76 dated 19 December 2013) and written informed consent, 18 patients undergoing surgery of the elbow, forearm, wrist, or hand were prospectively recruited based on the criteria below.

ELIGIBILITY:
Inclusion Criteria:

* patient's age between 18 and 80 years old,
* American Society of Anesthesiologists (ASA) physical status I - III,
* body mass index (BMI) between 20 and 35 kg/m2 and
* planned for surgery of the forearm, wrist, or hand.

Exclusion Criteria:

* patient's inability to give consent to the study,
* pre-existing neuropathy,
* infection at the site of puncture,
* coagulopathy, and
* allergy to amides local anaesthetics.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Success rate (ability to proceed with surgery without the need for intravenous narcotics, general anaesthesia, rescue blocks or local infiltration by the surgeon) | participants will be followed up throughout operation duration
  Success rate - was equivalent to surgical anesthesia, defined as the ability to proceed with surgery without the need for intravenous narcotics, general anaesthesia, rescue blocks or local infiltration by the surgeon
  The adequacy of block was determined during assessment of motor and sensory blockade at predetermined intervals, every 5 minutes until 30 minutes; Please refer to the study detailed description.

SECONDARY OUTCOMES:
Performance parameters | participants will be followed up throughout the procedure
  Imaging time (defined as the time interval between contact of the ultrasound probe with the patient and the acquisition of a satisfactory sonoanatomy - a complete round short-axis view of the axillary artery) Needling time (defined as the time interval between the start of the needle insertion and the end of local anaesthetic injection through the needle) Performance time (defined as the sum of imaging and needling times).
Safety aspects and potential complications as measured by incidence of paraesthesia, vascular puncture, Horner's syndrome, dyspnoea and symptoms suggestive of LA toxicity | participants will be followed up throughout procedure, during operation and 1 week after the operation (via phone call)
  The incidence of paraesthesia and vascular puncture was recorded if any. Horner's syndrome, dyspnoea and symptoms suggestive of local anaesthetic toxicity were routinely checked.
adequacy of block for tourniquet application | participants will be followed up throughout operation
  The incidence of tourniquet pain

CONTACTS AND LOCATIONS:
Overall Officials: Beh Zhi Yuen, MD, M.Anaes, Principal Investigator — Department of Anaesthesiology, Faculty of Medicine, Univeristy of Malaya

REFERENCES:
- [Background] References 1. Chin KJ, Perlas A, Chan VW, et al. Needle visualization in ultrasound guided regional anaesthesia: challenges and solutions. Reg Anesth Pain Med 2008; 33:532-544 2. Hebbard P and Royse C. Ultrasound guided posterior approach to the infraclavicular brachial plexus. Anaesthesia 2007; 62: 539 3. Levesque S, Dion N, Desgagne MC. Endpoint for successful, ultrasound-guided infraclavicular brachial plexus block. Can J Anaesth 2008; 55:308. 4. Tran DQH, Charghi R, Finlayson RJ. The 'Double Bubble' Sign for Successful Infraclavicular Brachial Plexus Blockade. Anesth Analg 2006; 103:1048-1049 5. Tran DQH, Bertini P, Zaouter C, et al. A Prospective, Randomized Comparison Between Single- and Double-Injection Ultrasound-Guided Infraclavicular Brachial Plexus Block. Reg Anesth Pain Med 2010; 35:16-21 6. Tran DQH, Munoz L, Zaouter C, et al. A prospective, randomized comparison between single- and double-injection ultrasound-guided supraclavicular brachial plexus block. Reg Anesth Pain Med 2009; 34:420-424. 7. Tran DQH, Russo G, Munoz L, et al. A prospective, randomized comparison between ultrasound-guided supraclavicular, infraclavicular and axillary brachial plexus blocks. Reg Anesth Pain Med 2009; 34:366-371
- [Derived] Beh ZY, Hasan MS, Lai HY, Kassim NM, Md Zin SR, Chin KF. Posterior parasagittal in-plane ultrasound-guided infraclavicular brachial plexus block-a case series. BMC Anesthesiol. 2015 Jul 21;15:105. doi: 10.1186/s12871-015-0090-0. PMID 26194896